CLINICAL TRIAL: NCT04431856
Title: CO-PARENT: COVID-19 - Parent Action in Response to Emotions and Needs for Treatment
Acronym: Co-PARENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Jill May Ehrenreich, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20200484
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Anxiety; Depression; Traumatic Stress Disorder
Keywords: COVID-19
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress Disorders, Traumatic; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Condition (Experimental): Participants in the Immediate Condition group will receive a total of 4 sessions of Unified Protocol for COVID-19 Parenting Stress (UP-COVID) intervention
  Interventions: Behavioral: Unified Protocol for COVID-19 Parenting Stress (UP-COVID)
- Delayed Condition (Active Comparator): Participants in the Delayed Condition group will receive the Self Help Guide (SHG) by the National Child Traumatic Stress Network (NCTSN). They will then receive the UP-COVID intervention following their week 6 assessment
  Interventions: Behavioral: Unified Protocol for COVID-19 Parenting Stress (UP-COVID); Behavioral: SHG

INTERVENTIONS:
Behavioral: Unified Protocol for COVID-19 Parenting Stress (UP-COVID) — UP-COVID is a group therapy session with each session lasting approximately 60-90 minutes. The sessions will focus on cognitive and behavioral strategies for managing their own distress, anxiety and sadness related to COVID-19, as well as, strategies related to parenting in the midst of the crisis.
Behavioral: SHG — Brochure that details techniques for coping with stress.
  Arms: Delayed Condition

SUMMARY:
The purpose of this research study is to collect information to better understand caregiver responses to COVID-19 stress and to help caregivers cope with these stressors.

ELIGIBILITY:
Inclusion Criteria:

* consent to participate via RedCap
* indicate a mild or greater elevation on screening measures of anxiety, depression and/or traumatic stress
* have a child between 6 and 13 years
* speak/read English or Spanish fluently

Exclusion Criteria:

* reported severe mental illness (e.g., bipolar disorder, schizophrenia, an intellectual disability, psychosis, alcohol use disorder, substance use disorder) or hospitalization for mental health concerns or suicide attempt.
* reported prior arrest for child endangerment, child abuse or child neglect, or prior investigation by the Florida Department of Children and Families (DCF)
* may be excluded if the severity of current mental illness is such that outpatient, weekly group treatment would be considered inappropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
Measure of Anxiety as assessed by the OASIS | week 6 and week 12
  The Overall Anxiety Severity and Impairment Scale (OASIS) is a 5 self-reported questionnaire evaluating the severity and functional impairment due to anxiety. The total score ranges from 0 (no anxiety) to 20 (severe anxiety).
Measure of Depression as assessed by the ODSIS | week 6 and week 12
  Overall Depression Severity and Impairment Scale (ODSIS) is a 5-item measure assessing the frequency and intensity of depressive symptoms. The total score ranges from 0-20 with the higher score indicating increased depression.
Measure of PTSD as assessed by the PCL-5 | week 6 and week 12
  PTSD Checklist (PCL-5) is a 20-item measure of PTSD symptoms in adults. Total score ranges from 0 to 80 with the higher score indicating higher PTSD symptoms.

SECONDARY OUTCOMES:
Measure of Parenting Overprotection/Overcontrol as assessed by the S-EMBU | week 6 and week 12
  The Egna Minnen Betraffande Uppfostran - Short Form (S-EMBU) is a 9-item measure that assesses parents' perception of their overprotection/control. Total scores ranging from 9 (low overcontrol) to 36 (high overcontrol).
Measure of Parenting Rejection as assessed by the S-EMBU | week 6 and week 12
  The Egna Minnen Betraffande Uppfostran - Short Form is a 7-item measure that assesses parents' perception of their rejection. Total score ranging from 7 (low rejection) to 28 (high rejection).
Measure of Parenting Emotional Warmth as assessed by the S-EMBU | week 6 and week 12
  The Egna Minnen Betraffande Uppfostran - Short Form is a 6-item measure that assesses parents' perception of their emotional warmth. Total scores ranging from 6 (low warmth) to 24 (high warmth).
Measure of Parent Accommodation for Child Anxiety as assessed by the FASA | week 6 and week 12
  The Family Accommodation Scale - Anxiety (FASA) is a 13-item measure that assesses parent's accommodation of their child's anxiety related behaviors. Total scores range from 0 (low accommodation) to 52 (high accommodation).

CONTACTS AND LOCATIONS:
Overall Officials: Jill Ehrenreich-May, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No